CLINICAL TRIAL: NCT04667000
Title: The Effect Of Forced Air Warming Used For Different Body Parts During Caseraen Section On Maternal Hypothermia, Shivering, Thermal Comfort, Apgar Score And Breastfeeding: Randomized Controlled Trial
Brief Title: The Effect of Forced Air Warming During Caseraen Section on Maternal Hypothermia: Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Cigdem Yucel (Unknown); Ozgur Ozyuncu (Unknown)
Responsible Party: Principal Investigator, Cansu Akdag Topal, Research Asistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KA-180051
Record Dates: First submitted 2020-03-12; First posted 2020-12-14 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2021-12

CONDITIONS: Cesarean Section Complications; Hypothermia
Keywords: hypothermia; nursing care; cesarean section
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Intervention Model Description: parallel group randomized controlled study
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- lower extremities (Experimental): the women's lower extremities will be heated with Forced Air Warming
  Interventions: Other: Forced Air Warming
- upper extremities (Experimental): the women's upper extremities will be heated with Forced Air Warming
  Interventions: Other: Forced Air Warming
- whole body (Experimental): the women's whole body will be heated with Forced Air Warming
  Interventions: Other: Forced Air Warming
- control group (No Intervention): there is no intervention for this group

INTERVENTIONS:
Other: Forced Air Warming — We will use Forced Air Warming for cesarean patient
  Arms: lower extremities; upper extremities; whole body

SUMMARY:
During the cesarean section; Hypothermia can be seen due to reasons such as anesthesia, premedication drugs, cold operating room environment, exposure of tissues and organs, and use of cold intravenous fluids. Hypothermia associated with cesarean may affect maternal and fetal health negatively. As a result of hypothermia, coagulopathy, infection, undesirable cardiac events that cause an increase in oxygen consumption, delay in postoperative recovery and wound healing, postoperative nausea and vomiting, chills and relief may be observed in the mother. Newborns born from hypothermic mothers have lower body temperature, pH and Apgar scores. It is important to evaluate all women in terms of risk factors in the preoperative period in the prevention of hypothermia and complications related to hypothermia. Prevention of hypothermia, which has negative effects on maternal and newborn health, is one of the risks that the nurse can address independently. Therefore, this research; In order to determine the effect of heating different body areas using compressed air heating technique during cesarean section on hypothermia, tremor, thermal comfort, postpartum comfort and maternal satisfaction, a parallel group was planned as a randomized controlled trial. The study is planned to be conducted in Hacettepe University Adult Hospital Gynecology and Obstetrics Department delivery room and obstetrics service. Research data, Introductory Information Form (Appendix 1), Obstetric and Postpartum Features Form (Appendix 2), Patient Monitoring Form (Appendix 3), Termal Comfort Perception Scale (Appendix 4), Shivering Level Diagnostic Form (Appendix 5), LATCH Breastfeeding The Diagnostic and Measurement Tool (Appendix 6) will be collected using the Visual Analogue Scale (Appendix 7) and the Thermal Comfort Scale that will be developed by the researchers. Pregnant women who meet the inclusion criteria will be included in the research. Women will be divided into 4 groups as the lower extremities are heated, the upper extremities are heated, the whole body is heated, and the control group. According to the group of women; It will be heated 30 minutes before surgery and 30 minutes after surgery with lower limb, upper limb or whole body. Women in the control group will not be heated.

DETAILED DESCRIPTION:
This study was planned as a parallel group randomized controlled study in order to determine the effect of heating different body parts using forced air warming technique during cesarean section on maternal hypothermia, shivering, thermal comfort, the Apgar score of the newborn and breastfeeding.

In the preparation phase of the research; Determining the rate of hypothermia in women applying to the delivery room of Hacettepe University Adult Hospital for planned cesarean section, determining and procuring the devices to be used in the study, and establishing experimental and control groups will be realized.

Body temperatures of women will be measured for 2 weeks in order to determine the rate of hypothermia in women who have had cesarean section in the institution where the study will be conducted. Body temperature of women will be started 30 minutes before the cesarean section and will be measured every 15 minutes until 30 minutes after the operation. By determining the prevalence of hypothermia after cesarean section in women; It is aimed to reveal the necessity of heating with compressed air heating technique.

* Women are admitted to the delivery room 60-90 minutes before the cesarean operation. The Introductory Information Form will be applied by the researcher using face-to-face interview before the women are admitted to the operating room.
* 30 minutes before the operation, women's body temperature, shivering, blood pressure, pulse and respiratory values will be evaluated every 15 minutes and recorded on the Patient Monitoring Form. In addition, the Temperature Comfort Scale, which will be developed by the researchers, will be applied by face to face interview method.

Applications During Cesarean Surgery

* During the operation, women's body temperature, temperature comfort score, shivering, blood pressure, pulse, respiration and SpO2 values will be evaluated every 15 minutes and recorded on the Patient Monitoring Form.
* With the birth of the baby; The newborn's body temperature, 1st and 5th minute Apgar score will be evaluated and recorded on the Obstetric and Postpartum Characteristics Form.

Applications to be Made Within 30 Minutes After Cesarean Surgery

* After the cesarean operation, women will be monitored in the recovery unit for 30 minutes. Body temperature, temperature comfort score, shivering, blood pressure, pulse, respiration and SpO2 values will be evaluated every 15 minutes after the women are admitted to the recovery unit and recorded on the Patient Monitoring Form. In addition, the Temperature Comfort Scale, which will be developed by the researchers, will be applied to women 30 minutes after the operation for the second time.
* The pain level of women will be evaluated with the Visual Pain Scale 30 minutes after surgery.
* In the institution where the research will be conducted, all women are given a heated blanket at 70 0C when they feel cold and shiver after cesarean section. The number of covers used varies depending on the demand of the woman. Researcher women will not interrupt this routine care they receive. The number of heated covers used by women will be recorded on the Obstetric and Postpartum Characteristics Form.

Applications to be Performed in Obstetrics and Gynecology Service after Cesarean Operation

* Information such as the need for analgesia, time to start breastfeeding, first mobilization time, gas, stool and urine output will be obtained from the patient file and recorded in the Obstetric and Postpartum Characteristics Form.
* The pain level of women will be evaluated repeatedly with the Visual Pain Scale (VAS) at the 24th hour after surgery. Due to the effect of anesthesia and the administration of analgesics upon the request of the doctor within the first day after cesarean operation, the VAS score after 24 hours will be evaluated.
* Before discharge, the development of postpartum complications in a woman will be evaluated and recorded on the Obstetric and Postpartum Features Form.
* At Hacettepe University Adult Hospital Gynecology Service, the breastfeeding status of mothers of newborns is evaluated using the LATCH Breastfeeding Diagnostic and Measurement Tool. Effective breastfeeding score assessed by the nurses: LACTH score will be evaluated and recorded on the Obstetric and Postpartum Characteristics Form.

ELIGIBILITY:
Inclusion Criteria:

* - between the ages of 18-35
* Speak, understand and write Turkish
* 37 weeks and more pregnant
* ASA I (Normal, a disease other than surgical pathology that does not cause a systemic disorder or a healthy person without a systemic problem)
* Spinal anesthesia is planned
* No high-risk pregnancy diagnosis (Oligodydroamniosis, early membrane rupture, gestational diabetes mellitus, preeclampsia, fetal tachycardia, nonreactive NST, intrauterine growth retardation)
* Body mass index> 19 kg / m2 and <40 kg / m2,
* Having a single pregnancy and
* Pregnant women who agreed to participate in the study will be included in the sample.

Exclusion Criteria:

* - Emergency cesarean section
* Individuals with Forced Air Warming contraindications (Acute infection, Maternal fever before operation, etc.)
* In case of any complication that may develop in the mother or newborn at any stage of the research
* Pregnant women who want to leave the research at any stage of the research will be excluded from the sample.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Maternal Hypothermia | 30 minutes before the intervention to 30 minutes after the intervention.
  Maternal hypothermia is defined as body temperature falling below 36 ° C.

SECONDARY OUTCOMES:
Shivering | 30 minutes before the intervention to 30 minutes after the intervention.
  Shivering is a bodily function in response to cold in humans
Thermal Comfort | 30 minutes before the intervention to 30 minutes after the intervention.
  Thermal comfort is defined as the condition of mind that expresses satisfaction with the thermal environment.
Apgar Score | 30 minutes before the intervention to 30 minutes after the intervention.
  An objective score of the condition of a baby after birth. This score is determined by scoring the heart rate, respiratory effort, muscle tone, skin color, and response to a catheter in the nostril.
Breastfeeding Timing | 30 minutes before the intervention to 30 minutes after the intervention.
  The time between the start of breastfeeding of the newborn after birth

CONTACTS AND LOCATIONS:
Overall Officials: Ozgur Ozyuncu, PhD, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akhtar Z, Hesler BD, Fiffick AN, Mascha EJ, Sessler DI, Kurz A, Ayad S, Saager L. A randomized trial of prewarming on patient satisfaction and thermal comfort in outpatient surgery. J Clin Anesth. 2016 Sep;33:376-85. doi: 10.1016/j.jclinane.2016.04.041. Epub 2016 Jun 3. PMID 27555196
- [Background] Apfelbaum JL, Silverstein JH, Chung FF, Connis RT, Fillmore RB, Hunt SE, Nickinovich DG, Schreiner MS, Silverstein JH, Apfelbaum JL, Barlow JC, Chung FF, Connis RT, Fillmore RB, Hunt SE, Joas TA, Nickinovich DG, Schreiner MS; American Society of Anesthesiologists Task Force on Postanesthetic Care. Practice guidelines for postanesthetic care: an updated report by the American Society of Anesthesiologists Task Force on Postanesthetic Care. Anesthesiology. 2013 Feb;118(2):291-307. doi: 10.1097/ALN.0b013e31827773e9. No abstract available. PMID 23364567
- [Background] Arkilic CF, Akca O, Taguchi A, Sessler DI, Kurz A. Temperature monitoring and management during neuraxial anesthesia: an observational study. Anesth Analg. 2000 Sep;91(3):662-6. doi: 10.1097/00000539-200009000-00031. PMID 10960396
- [Background] Badjatia N, Strongilis E, Gordon E, Prescutti M, Fernandez L, Fernandez A, Buitrago M, Schmidt JM, Ostapkovich ND, Mayer SA. Metabolic impact of shivering during therapeutic temperature modulation: the Bedside Shivering Assessment Scale. Stroke. 2008 Dec;39(12):3242-7. doi: 10.1161/STROKEAHA.108.523654. Epub 2008 Oct 16. PMID 18927450
- [Background] Bender M, Self B, Schroeder E, Giap B. Comparing new-technology passive warming versus traditional passive warming methods for optimizing perioperative body core temperature. AORN J. 2015 Aug;102(2):183.e1-8. doi: 10.1016/j.aorn.2015.06.005. PMID 26227528
- [Background] Betran AP, Ye J, Moller AB, Zhang J, Gulmezoglu AM, Torloni MR. The Increasing Trend in Caesarean Section Rates: Global, Regional and National Estimates: 1990-2014. PLoS One. 2016 Feb 5;11(2):e0148343. doi: 10.1371/journal.pone.0148343. eCollection 2016. PMID 26849801
- [Background] Carpenter L, Baysinger CL. Maintaining perioperative normothermia in the patient undergoing cesarean delivery. Obstet Gynecol Surv. 2012 Jul;67(7):436-46. doi: 10.1097/OGX.0b013e3182605ccd. PMID 22926250
- [Background] Chakladar A, Dixon MJ, Crook D, Harper CM. The effects of a resistive warming mattress during caesarean section: a randomised, controlled trial. Int J Obstet Anesth. 2014 Nov;23(4):309-16. doi: 10.1016/j.ijoa.2014.06.003. Epub 2014 Jun 13. PMID 25266313
- [Background] Chebbout R, Newton RS, Walters M, Wrench IJ, Woolnough M. Does the addition of active body warming to in-line intravenous fluid warming prevent maternal hypothermia during elective caesarean section? A randomised controlled trial. Int J Obstet Anesth. 2017 May;31:37-44. doi: 10.1016/j.ijoa.2017.04.008. Epub 2017 Apr 27. PMID 28576354
- [Background] Chung SH, Lee BS, Yang HJ, Kweon KS, Kim HH, Song J, Shin DW. Effect of preoperative warming during cesarean section under spinal anesthesia. Korean J Anesthesiol. 2012 May;62(5):454-60. doi: 10.4097/kjae.2012.62.5.454. Epub 2012 May 24. PMID 22679543
- [Background] Cobb B, Cho Y, Hilton G, Ting V, Carvalho B. Active Warming Utilizing Combined IV Fluid and Forced-Air Warming Decreases Hypothermia and Improves Maternal Comfort During Cesarean Delivery: A Randomized Control Trial. Anesth Analg. 2016 May;122(5):1490-7. doi: 10.1213/ANE.0000000000001181. PMID 26895002
- [Background] Duff J, Di Staso R, Cobbe KA, Draper N, Tan S, Halliday E, Middleton S, Lam L, Walker K. Preventing hypothermia in elective arthroscopic shoulder surgery patients: a protocol for a randomised controlled trial. BMC Surg. 2012 Jul 20;12:14. doi: 10.1186/1471-2482-12-14. PMID 22817672
- [Background] Fallis WM, Hamelin K, Symonds J, Wang X. Maternal and newborn outcomes related to maternal warming during cesarean delivery. J Obstet Gynecol Neonatal Nurs. 2006 May-Jun;35(3):324-31. doi: 10.1111/j.1552-6909.2006.00052.x. PMID 16700681
- [Background] Geller EJ, Wu JM, Jannelli ML, Nguyen TV, Visco AG. Maternal outcomes associated with planned vaginal versus planned primary cesarean delivery. Am J Perinatol. 2010 Oct;27(9):675-83. doi: 10.1055/s-0030-1249765. Epub 2010 Mar 16. PMID 20235001
- [Background] Haas DM, Morgan S, Contreras K, Enders S. Vaginal preparation with antiseptic solution before cesarean section for preventing postoperative infections. Cochrane Database Syst Rev. 2018 Jul 17;7(7):CD007892. doi: 10.1002/14651858.CD007892.pub6. PMID 30016540
- [Background] Harper CM, Andrzejowski JC, Alexander R. NICE and warm. Br J Anaesth. 2008 Sep;101(3):293-5. doi: 10.1093/bja/aen233. No abstract available. PMID 18710834
- [Background] Hess PE, Snowman CE, Wang J. Hypothermia after cesarean delivery and its reversal with lorazepam. Int J Obstet Anesth. 2005 Oct;14(4):279-83. doi: 10.1016/j.ijoa.2005.02.004. PMID 16143507
- [Background] Horn EP, Bein B, Steinfath M, Ramaker K, Buchloh B, Hocker J. The incidence and prevention of hypothermia in newborn bonding after cesarean delivery: a randomized controlled trial. Anesth Analg. 2014 May;118(5):997-1002. doi: 10.1213/ANE.0000000000000160. PMID 24681658
- [Background] Horn EP, Schroeder F, Gottschalk A, Sessler DI, Hiltmeyer N, Standl T, Schulte am Esch J. Active warming during cesarean delivery. Anesth Analg. 2002 Feb;94(2):409-14, table of contents. doi: 10.1097/00000539-200202000-00034. PMID 11812709
- [Background] Jaiyeoba O. Postoperative infections in obstetrics and gynecology. Clin Obstet Gynecol. 2012 Dec;55(4):904-13. doi: 10.1097/GRF.0b013e3182714734. PMID 23090459
- [Background] Jensen D, Wallace S, Kelsay P. LATCH: a breastfeeding charting system and documentation tool. J Obstet Gynecol Neonatal Nurs. 1994 Jan;23(1):27-32. doi: 10.1111/j.1552-6909.1994.tb01847.x. PMID 8176525
- [Background] John M, Ford J, Harper M. Peri-operative warming devices: performance and clinical application. Anaesthesia. 2014 Jun;69(6):623-38. doi: 10.1111/anae.12626. Epub 2014 Apr 10. PMID 24720346
- [Background] Kurz A. Thermal care in the perioperative period. Best Pract Res Clin Anaesthesiol. 2008 Mar;22(1):39-62. doi: 10.1016/j.bpa.2007.10.004. PMID 18494388
- [Background] Kurz A. Physiology of thermoregulation. Best Pract Res Clin Anaesthesiol. 2008 Dec;22(4):627-44. doi: 10.1016/j.bpa.2008.06.004. PMID 19137807
- [Background] Leeth D, Mamaril M, Oman KS, Krumbach B. Normothermia and patient comfort: a comparative study in an outpatient surgery setting. J Perianesth Nurs. 2010 Jun;25(3):146-51. doi: 10.1016/j.jopan.2010.03.010. PMID 20511085
- [Background] Letko MD. Understanding the Apgar score. J Obstet Gynecol Neonatal Nurs. 1996 May;25(4):299-303. doi: 10.1111/j.1552-6909.1996.tb02575.x. PMID 8708830
- [Background] May T, Seder DB, Fraser GL, Tu C, McCrum B, Lucas L, Riker RR. Association of the Bedside Shivering Assessment Scale and derived EMG power during therapeutic hypothermia in survivors of cardiac arrest. Resuscitation. 2011 Aug;82(8):1100-3. doi: 10.1016/j.resuscitation.2011.03.037. Epub 2011 Apr 16. PMID 21592643
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG; Consolidated Standards of Reporting Trials Group. CONSORT 2010 Explanation and Elaboration: Updated guidelines for reporting parallel group randomised trials. J Clin Epidemiol. 2010 Aug;63(8):e1-37. doi: 10.1016/j.jclinepi.2010.03.004. Epub 2010 Mar 25. PMID 20346624
- [Background] Mpogoro FJ, Mshana SE, Mirambo MM, Kidenya BR, Gumodoka B, Imirzalioglu C. Incidence and predictors of surgical site infections following caesarean sections at Bugando Medical Centre, Mwanza, Tanzania. Antimicrob Resist Infect Control. 2014 Aug 11;3:25. doi: 10.1186/2047-2994-3-25. eCollection 2014. PMID 25126415
- [Background] Mylonas I, Friese K. Indications for and Risks of Elective Cesarean Section. Dtsch Arztebl Int. 2015 Jul 20;112(29-30):489-95. doi: 10.3238/arztebl.2015.0489. PMID 26249251
- [Background] Ng SF, Oo CS, Loh KH, Lim PY, Chan YH, Ong BC. A comparative study of three warming interventions to determine the most effective in maintaining perioperative normothermia. Anesth Analg. 2003 Jan;96(1):171-6, table of contents. doi: 10.1097/00000539-200301000-00036. PMID 12505947
- [Background] Paris LG, Seitz M, McElroy KG, Regan M. A randomized controlled trial to improve outcomes utilizing various warming techniques during cesarean birth. J Obstet Gynecol Neonatal Nurs. 2014 Nov-Dec;43(6):719-28. doi: 10.1111/1552-6909.12510. Epub 2014 Oct 14. PMID 25316112
- [Background] Price DD, McGrath PA, Rafii A, Buckingham B. The validation of visual analogue scales as ratio scale measures for chronic and experimental pain. Pain. 1983 Sep;17(1):45-56. doi: 10.1016/0304-3959(83)90126-4. PMID 6226917
- [Background] Rajagopalan S, Mascha E, Na J, Sessler DI. The effects of mild perioperative hypothermia on blood loss and transfusion requirement. Anesthesiology. 2008 Jan;108(1):71-7. doi: 10.1097/01.anes.0000296719.73450.52. PMID 18156884
- [Background] Scott EM, Buckland R. A systematic review of intraoperative warming to prevent postoperative complications. AORN J. 2006 May;83(5):1090-104, 1107-13. doi: 10.1016/s0001-2092(06)60120-8. PMID 16722286
- [Background] Sessler DI. Complications and treatment of mild hypothermia. Anesthesiology. 2001 Aug;95(2):531-43. doi: 10.1097/00000542-200108000-00040. No abstract available. PMID 11506130
- [Background] Sessler DI. Perioperative heat balance. Anesthesiology. 2000 Feb;92(2):578-96. doi: 10.1097/00000542-200002000-00042. PMID 10691247
- [Background] Smaill FM, Grivell RM. Antibiotic prophylaxis versus no prophylaxis for preventing infection after cesarean section. Cochrane Database Syst Rev. 2014 Oct 28;2014(10):CD007482. doi: 10.1002/14651858.CD007482.pub3. PMID 25350672
- [Background] Sultan P, Habib AS, Cho Y, Carvalho B. The Effect of patient warming during Caesarean delivery on maternal and neonatal outcomes: a meta-analysis. Br J Anaesth. 2015 Oct;115(4):500-10. doi: 10.1093/bja/aev325. PMID 26385660
- [Background] Sahin A, Aypar U. Effect of amino acid solutions on intraoperative hypothermia and postoperative shivering. Comparison of two anesthetic regimens. Acta Anaesthesiol Scand. 2002 Jan;46(1):64-7. PMID 11903074
- [Background] Torloni MR, Betran AP, Souza JP, Widmer M, Allen T, Gulmezoglu M, Merialdi M. Classifications for cesarean section: a systematic review. PLoS One. 2011 Jan 20;6(1):e14566. doi: 10.1371/journal.pone.0014566. PMID 21283801
- [Background] Wagner D, Byrne M, Kolcaba K. Effects of comfort warming on preoperative patients. AORN J. 2006 Sep;84(3):427-48. doi: 10.1016/s0001-2092(06)63920-3. PMID 17004666
- [Background] Warttig S, Alderson P, Campbell G, Smith AF. Interventions for treating inadvertent postoperative hypothermia. Cochrane Database Syst Rev. 2014 Nov 20;2014(11):CD009892. doi: 10.1002/14651858.CD009892.pub2. PMID 25411963
- [Background] Woolnough M, Allam J, Hemingway C, Cox M, Yentis SM. Intra-operative fluid warming in elective caesarean section: a blinded randomised controlled trial. Int J Obstet Anesth. 2009 Oct;18(4):346-51. doi: 10.1016/j.ijoa.2009.02.009. Epub 2009 Aug 7. PMID 19665366
- [Background] Wu X. The safe and efficient use of forced-air warming systems. AORN J. 2013 Mar;97(3):302-8. doi: 10.1016/j.aorn.2012.12.008. PMID 23452695
- [Background] Yokoyama K, Suzuki M, Shimada Y, Matsushima T, Bito H, Sakamoto A. Effect of administration of pre-warmed intravenous fluids on the frequency of hypothermia following spinal anesthesia for Cesarean delivery. J Clin Anesth. 2009 Jun;21(4):242-8. doi: 10.1016/j.jclinane.2008.12.010. Epub 2009 Jun 6. PMID 19502035